CLINICAL TRIAL: NCT01516541
Title: A Phase 3b, Multi-Center, Double-Blind, Placebo-Controlled, Parallel Group, Study to Evaluate the Effect of Dalcetrapib 600 mg on Cardiovascular (CV) Events in Adult Patients With Stable Coronary Heart Disease (CHD), CHD Risk Equivalents or at Elevated Risk for Cardiovascular Disease (CVD).
Brief Title: A Study of Dalcetrapib in Patients With Stable Coronary Heart Disease, With Coronary Heart Disease Risk Equivalents or at Elevated Risk for Cardiovascular Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NC25608; 2011-001891-21 (EudraCT Number)
Record Dates: First submitted 2012-01-13; First posted 2012-01-25 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Cardiovascular Disease, Coronary Heart Disease, Dyslipidemia, Peripheral Arterial Disease (PAD)
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Dyslipidemias; Peripheral Arterial Disease | interventions — dalcetrapib

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Dalcetrapib (Experimental): Dalcetrapib 600 mg orally daily on a background of contemporary, guidelines-based medical care.
  Interventions: Other: Background care; Drug: dalcetrapib
- Placebo (Placebo Comparator): Placebo orally daily, on a background of contemporary, guidelines-based medical care.
  Interventions: Other: Background care; Drug: Placebo

INTERVENTIONS:
Other: Background care — Guidelines-based medical care
Drug: Placebo — Matching dalcetrapib placebo orally daily
  Arms: Placebo
Drug: dalcetrapib — 600 mg orally daily
  Arms: Dalcetrapib

SUMMARY:
This multicenter, randomized, double-blind, placebo-controlled, parallel-group study will evaluate the potential of dalcetrapib to reduce cardiovascular morbidity and mortality in patients with stable coronary heart disease (CHD), with CHD risk equivalents or at elevated risk for cardiovascular disease. Eligible patients will be randomized to receive either dalcetrapib 600 mg orally daily or placebo orally daily, on a background of contemporary, guidelines-based medical care. Anticipated time on study treatment is 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 45 years of age
* Established cardiovascular disease A stable coronary disease B cerebrovascular disease C peripheral artery disease
* Without established coronary disease D pharmacologically treated type 2 diabetes mellitus and one or more risk factor(s) for cardiovascular disease E 3 or more risk factors for cardiovascular disease
* Receiving evidence-based medical and dietary management of dyslipidemia

Exclusion Criteria:

* Occurrence of myocardial infarction, hospitalization for unstable angina, stroke or revascularization (coronary, carotid or peripheral) within three months prior to randomization
* Uncontrolled hypertension
* Uncontrolled diabetes
* Concomitant treatment with any other drug raising HDL-C
* Previous treatment with compounds targeting cholesteryl ester transfer protein (CETP)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2220 (Actual)
Dates: Start 2012-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Time to first occurrence of any component of the composite cardiovascular event (cardiovascular mortality and morbidity) | approximately 4 years

SECONDARY OUTCOMES:
All cause mortality | approximately 4 years
Safety: Incidence of adverse events | approximately 4 years
Change in blood lipid and lipoprotein levels | from baseline to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (217):
- United States (115):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Anaheim, California
  - Fullerton, California
  - San Diego, California
  - Santa Ana, California
  - Santa Rosa, California
  - Torrance, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Lonetree, Colorado
  - Bridgeport, Connecticut
  - Hartford, Connecticut
  - Boynton Beach, Florida
  - Daytona Beach, Florida
  - Fort Myers, Florida
  - Jacksonville, Florida
  - Panama City, Florida
  - Plantation, Florida
  - Port Charlotte, Florida
  - Tallahassee, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Covington, Georgia
  - Cumming, Georgia
  - Decatur, Georgia
  - Aurora, Illinois
  - Rock Island, Illinois
  - Winfield, Illinois
  - Elkhart, Indiana
  - Hammond, Indiana
  - Indianapolis, Indiana
  - Muncie, Indiana
  - South Bend, Indiana
  - Overland Park, Kansas
  - Louisville, Kentucky
  - Alexandria, Louisiana
  - Bangor, Maine
  - Beltsville, Maryland
  - Salisbury, Maryland
  - Boston, Massachusetts
  - Haverhill, Massachusetts
  - Hyannis, Massachusetts
  - North Dartmouth, Massachusetts
  - Jackson, Michigan
  - Kalamazoo, Michigan
  - Marquette, Michigan
  - Midland, Michigan
  - Rochester Hills, Michigan
  - Saginaw, Michigan
  - Ypsilanti, Michigan
  - Rochester, Minnesota
  - Saint Cloud, Minnesota
  - Chesterfield, Missouri
  - Columbia, Missouri
  - Kansas City, Missouri
  - Kalispell, Montana
  - Nashua, New Hampshire
  - Camden, New Jersey
  - Haddon Heights, New Jersey
  - Mine Hill, New Jersey
  - Wayne, New Jersey
  - Westwood, New Jersey
  - Albany, New York
  - Buffalo, New York
  - Cortlandt Manor, New York
  - Poughkeepsi, New York
  - Saratoga Springs, New York
  - Smithtown, New York
  - Syracuse, New York
  - The Bronx, New York
  - Troy, New York
  - Asheville, North Carolina
  - Durham, North Carolina
  - Elizabeth City, North Carolina
  - Hickory, North Carolina
  - Morehead City, North Carolina
  - Rocky Mount, North Carolina
  - Statesville, North Carolina
  - Wilmington, North Carolina
  - Fargo, North Dakota
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Mansfield, Ohio
  - Mentor, Ohio
  - Thornville, Ohio
  - Toledo, Ohio
  - Zanesville, Ohio
  - Allentowm, Pennsylvania
  - Altoona, Pennsylvania
  - Camp Hill, Pennsylvania
  - Doylestown, Pennsylvania
  - Erie, Pennsylvania
  - Langhorne, Pennsylvania
  - Lansdale, Pennsylvania
  - North Wales, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pottstown, Pennsylvania
  - Tipton, Pennsylvania
  - West Chester, Pennsylvania
  - Anderson, South Carolina
  - Greer, South Carolina
  - Rapid City, South Dakota
  - Johnson City, Tennessee
  - Dallas, Texas
  - Humble, Texas
  - Odessa, Texas
  - Tyler, Texas
  - Provo, Utah
  - Charlottesville, Virginia
  - Danville, Virginia
  - Lynchburg, Virginia
  - Manassas, Virginia
  - Richmond, Virginia
  - Winchester, Virginia
- Australia (3):
  - Milton, Queensland
  - Geelong, Victoria
  - Joondalup, Western Australia
- Canada (24):
  - Coquitlam, British Columbia
  - Kelowna, British Columbia
  - Vancouver, British Columbia
  - Moncton, New Brunswick
  - Ajax, Ontario
  - Barrie, Ontario
  - Burlington, Ontario
  - Cambridge, Ontario
  - Greater Sudbury, Ontario
  - London, Ontario
  - Oakville, Ontario
  - Oshawa, Ontario
  - Thunder Bay, Ontario
  - Toronto, Ontario
  - Granby, Quebec
  - Greenfield Park, Quebec
  - Lachine, Quebec
  - Longueuil, Quebec
  - Mirabel, Quebec
  - Montreal, Quebec
  - Québec, Quebec
  - Saint-Lambert, Quebec
  - Trois-Rivières, Quebec
  - Val-d'Or, Quebec
- China (3):
  - Beijing
  - Nanchang
  - Shijiazhuang
- Czechia (7):
  - Benátky nad Jizerou
  - Jindřichův Hradec
  - Ostrava
  - Pardubice
  - Prague
  - Slaný
  - Trutnov
- Denmark (4):
  - Århus N
  - Ballerup Municipality
  - Hvidovre
  - Vejle
- Pessac, France
- Hungary (7):
  - Budapest
  - Debrecen
  - Kisvárda
  - Komárom
  - Nagykanizsa
  - Pécs
  - Úrhida
- Mexico (16):
  - Aguascalientes
  - Aguascaliente
  - Celaya
  - Chihuahua City
  - Cuernavaca
  - D. F.
  - Durango
  - Guadalajara
  - Mexico City
  - Monterrey
  - Pachuca
  - Querétaro
  - San Luis Potosi S.l.p.
  - San Luis Potosí City
  - San Luís Potosí
  - Tampico
- Netherlands (16):
  - Alkmaar
  - Amsterdam
  - Apeldoorn
  - Breda
  - Delft
  - Eindhoven
  - Gouda
  - Groningen
  - Heerlen
  - Hoorn
  - Leiden
  - Rotterdam
  - Utrecht
  - Velp
  - Venlo
  - Zoetermeer
- Poland (11):
  - Bialystok
  - Gdansk
  - Gdynia
  - Katowice
  - Krakow
  - Lodz
  - Lublin
  - Poznan
  - Pulway
  - Ruda Śląska
  - Warsaw
- Spain (4):
  - Almería, Almeria
  - Barcelona, Barcelona
  - Madrid, Madrid
  - Málaga, Malaga
- United Kingdom (6):
  - Birmingham
  - Cardiff
  - Glasgow
  - Liverpool
  - Manchester
  - Reading